CLINICAL TRIAL: NCT00478361
Title: A Phase II Study of Gemcitabine, Paclitaxel, and Doxorubicin, With Pegfilgrastim for the Treatment of Patients With Metastatic Transitional Cell Carcinoma and Renal Insufficiency
Brief Title: Gemcitabine, Paclitaxel, Doxorubicin in Metastatic or Unresectable Bladder Cancer With Decreased Kidney Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0839; NCI-2009-00154 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000544831; 2U10CA045809-17 (NIH); NCT00477438 (obsolete NCT alias)
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-09

CONDITIONS: Distal Urethral Cancer; Metastatic Transitional Cell Cancer of the Renal Pelvis and Ureter; Proximal Urethral Cancer; Recurrent Bladder Cancer; Recurrent Transitional Cell Cancer of the Renal Pelvis and Ureter; Recurrent Urethral Cancer; Regional Transitional Cell Cancer of the Renal Pelvis and Ureter; Stage III Bladder Cancer; Stage IV Bladder Cancer; Transitional Cell Carcinoma of the Bladder; Urethral Cancer Associated With Invasive Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Gemcitabine; Paclitaxel; Taxes; Doxorubicin; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine, Paclitaxel and Doxorubicin (Experimental): Paclitaxel 135 mg/m^2 intravenous (IV) over 1 hour; Gemcitabine 900 mg/m^2 IV over 90 min; Doxorubicin 40 mg/m^2 IV over 20 min; treatment may repeat every 2 weeks for up to nine courses. Injection of Pegfilgrastim on day 1.
  Interventions: Drug: Gemcitabine hydrochloride; Drug: Paclitaxel; Drug: Doxorubicin hydrochloride; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Gemcitabine hydrochloride — Gemcitabine 900 mg/m^2 IV over 90 minutes repeat every 14 days.
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: Paclitaxel — 135 mg/m^2 IV over 1 hour
  Other Names: Anzatax; Asotax; TAX; Taxol
Drug: Doxorubicin hydrochloride — Doxorubicin 40 mg/m^2 IV over 20 minutes
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: Pegfilgrastim — Subcutaneously injection on day 1.
  Other Names: Filgrastim SD-01; GCSF-SD01; Neulasta; SD-01 sustained duration G-CSF

SUMMARY:
This phase II trial is studying how well giving gemcitabine, paclitaxel, and doxorubicin together with pegfilgrastim works in treating patients with metastatic or unresectable bladder cancer or urinary tract cancer and kidney dysfunction. Drugs used in chemotherapy, such as gemcitabine, paclitaxel, and doxorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Colony stimulating factors, such as pegfilgrastim, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy. Giving combination chemotherapy together with pegfilgrastim may kill more tumor cells. Chemotherapy drugs may have different effects in patients who have changes in their kidney function.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the efficacy of gemcitabine hydrochloride, paclitaxel, doxorubicin hydrochloride, and pegfilgrastim, in terms of response rate, in patients with metastatic or unresectable transitional cell carcinoma of the bladder or urinary tract and renal insufficiency.

SECONDARY OBJECTIVES:

I. Assess the safety and tolerability of this regimen in these patients. II. Determine the median time to progression in patients treated with this regimen.

III. Determine the median survival duration in patients treated with this regimen.

IV. Assess the safety and efficacy of pegfilgrastim in these patients.

OUTLINE: This is a multicenter study.

Patients receive doxorubicin hydrochloride intravenous (IV) over 20 minutes, paclitaxel IV over 60 minutes, gemcitabine hydrochloride IV over 90 minutes, and pegfilgrastim subcutaneously on day 1. Treatment repeats every 14 days for up to 9 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed transitional cell carcinoma (TCC) of the bladder, urethra, or upper urinary tract
* Mixed TCC and variant histologies (i.e., small cell, squamous cell, adenocarcinoma, or sarcoma) allowed if present in < 50% of the biopsy specimen
* Patients must sign an informed consent indicating that they are aware of the investigational nature of this study, in keeping with the policies of the institution.
* Measurable disease: may include radiographic detection of metastases in lymph nodes (>= 1.5 cm) or liver or lung (>= 1.0 cm) OR pelvic mass palpable on examination under anesthesia
* Creatinine clearance < 60 mL/min; no renal insufficiency that requires hemodialysis; no renal insufficiency that is reversible in patients with tumor confined to the primary site (i.e., that is potentially resectable with neoadjuvant chemotherapy)
* Zubrod performance status 0-2
* Platelet count > 100,000/mm^3
* Absolute granulocyte count > 1,500/mm^3
* Bilirubin =< 2.0 mg/dL
* Aminotransferases (AST and ALT) =< 2 times upper limit of normal
* Left ventricular ejection fraction (LVEF) > 40% OR normal electrocardiogram (EKG or ECG) and no history of cardiac disease
* All patients must be evaluated in the Department of Genitourinary Medical Oncology at M. D. Anderson Cancer Center or participating CCOP center prior to signing informed consent.
* No prior systemic chemotherapy including, adjuvant or neoadjuvant therapy
* Prior intravesicular chemotherapy allowed

Exclusion Criteria:

* No brain metastases
* Not pregnant or nursing
* No severe or uncontrolled infection
* No New York Heart Association class III-IV congestive heart failure, unstable angina, or history of myocardial infarction within the past 6 months
* No peripheral neuropathy >= grade 2
* No persistently uncontrolled diabetes mellitus
* No chronic liver disease
* No HIV positivity
* No other malignancy except nonmelanoma skin cancer unless disease-free for the past 3 years
* No overt psychosis, mental disability, or other condition that would preclude giving informed consent
* No known sickle cell disease
* No uncontrolled severe hypertension
* Renal insufficiency that requires hemodialysis or renal insufficiency that is reversible in patients with tumor confined to the primary site (i.e., that is potentially resectable with neoadjuvant chemotherapy).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lance Pagliaro, MD, BA, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Ozark Health Ventures LLC dba Cancer Research for The Ozarks Springfield, Springfield, Missouri
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: April 24, 2007 to November 10, 2011. All recruitment done within Community Clinical Oncology Programs (CCOP) medical clinics, specifically The University of Texas MD Anderson Cancer Center and the Ozarks Regional CCOP.
Pre-assignment Details: One patient withdrew from the study without receiving treatment.
Groups:
- Gemcitabine, Paclitaxel and Doxorubicin: Paclitaxel 135 mg/m^2 intravenous (IV) over 1 hour; Gemcitabine 900 mg/m^2 IV over 90 minutes; Doxorubicin 40 mg/m^2 IV over 20 minutes; treatment may repeat every 2 weeks for up to nine courses. Subcutaneous Injection of Pegfilgrastim on day 1 or 2 of each course, after chemotherapy.
Period: Overall Study
Arm/Group | Gemcitabine, Paclitaxel and Doxorubicin
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine, Paclitaxel and Doxorubicin
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 72 [51 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The percentage of participants with either Complete Response (CR) or Partial Response (PR) in their disease burden based upon the rules of the Response Evaluation Criteria in Solid Tumors (RECIST). A participant with of all of the lesions disappearing is a CR. A participant with at least a 30 percent decrease in the measured lesions is a PR.
Time Frame: Up to 12 weeks, or following completion 6 cycles of chemotherapy, respectively; the best response achieved within 6 cycles of starting chemotherapy used to calculate response rate.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine, Paclitaxel and Doxorubicin
Number analyzed (Participants) | 39
percentage of participants | 56.4 [39.6 to 72.2]

2. Secondary Outcome: Overall Survival (OS) of Participants With a Continuous Complete Response, Partial Response and Stable Disease
Description: The overall survival was determined by grouping participants based upon their response based on RECIST. The groups are Complete Response(CR): All the cancerous lesion disappear, Partial Response (PR): All the measured lesions decrease by at least 30 percent, and Stable Disease(SD): No significant change in the disease burden. OS of complete response or partial response participants were compared to the reference group of stable disease participants in a Hazard Ratio(HR). If HR is greater than 1, the experimental group has a better outcome than the reference group. If HR is less than 1, the reference group has the better outcome.
Time Frame: Registration Date of each participant for up to three years or death whichever came first
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Gemcitabine, Paclitaxel and Doxorubicin
Number analyzed (Participants) | 39
Hazard Ratio
  Complete Response | 0.25 [0.07 to 0.95]
  Partial Response | 1.09 [0.44 to 2.70]

3. Secondary Outcome: Safety and Efficacy of Same-day Pegfilgrastim
Description: Determined the number of participants who had either a fever due to abnormally low level of neutrophils, a type of white blood cell, on the day of study drug treatment, or the participants who had the study drug treatment delayed due to an abnormally low level of neutrophils.
Time Frame: Up to 3 years
Population: Thirty-two patients (82%) received Pegfilgrastim immediately after chemotherapy on day 1 of the cycle.
Measure: Number; unit: participants
Arm/Group | Gemcitabine, Paclitaxel and Doxorubicin
Number analyzed (Participants) | 32
participants
  Neutropenic Fever | 4
  Treatment Delay | 0

ADVERSE EVENTS:
Time Frame: Adverse event collection during therapy may continue for 12 weeks (6 cycles) with possible 3 additional cycles (6 weeks) beyond a documented complete response.
Description: AEs were graded by numerical score according to the NCI Common Terminology Criteria Adverse Events (CTCAE), version 4.0.
Arm/Group | Gemcitabine, Paclitaxel and Doxorubicin
Serious Adverse Events (participants affected / at risk) | 39/39
Other Adverse Events (participants affected / at risk) | 34/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Paclitaxel and Doxorubicin (N=39)
Granulocytopenia (Blood and lymphatic system disorders) | 13 (13)
Lymphopenia (Investigations) | 3 (3)
Leukopenia (Investigations) | 8 (8)
Anemia (Blood and lymphatic system disorders) | 6 (6)
Thrombocytopenia (Investigations) | 6 (6)
Neutropenic Fever (Blood and lymphatic system disorders) | 4 (4)
Fatigue (General disorders) | 4 (4)
Hyperuricemia (Metabolism and nutrition disorders) | 4 (4)
Mucositis (Gastrointestinal disorders) | 4 (4)
Deep Vein Thrombosis (Vascular disorders) | 2 (2)
Pain (General disorders) | 3 (3)
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 (2)
Hand Foot Syndrome (Musculoskeletal and connective tissue disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Paclitaxel and Doxorubicin (N=39)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (6)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Platelet Count Decreased (Investigations) | 13 (28)
Anemia (Blood and lymphatic system disorders) | 32 (73)
Fever (General disorders) | 3 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 10 (10)
Skin and Subcutaneous Tissue Disorders - Nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Creatinine Increased (Investigations) | 26 (38)
Hyperglycemia (Metabolism and nutrition disorders) | 14 (18)
Peripheral Motor Neuropathy (Nervous system disorders) | 2 (2)
Skin and Subcutaneous Tissue Disorders - Redness/Irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Edema Limbs (General disorders) | 10 (12)
Alkaline Phosphatase Increased (Investigations) | 6 (8)
Peripheral Sensory Neuropathy (Nervous system disorders) | 13 (17)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
BUN (Blood and lymphatic system disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2)
Mucositis Oral (Gastrointestinal disorders) | 8 (14)
Carbon Monoxide Diffusing Capacity Decreased (Investigations) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (12)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Cardiac Troponin I Increased (Investigations) | 1 (2)
Watering Eyes (Eye disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 4 (5)
Fatigue (General disorders) | 17 (33)
Anorexia (Metabolism and nutrition disorders) | 11 (14)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (6)
Hematuria (Renal and urinary disorders) | 6 (8)
White Blood Cell Decreased (Investigations) | 5 (8)
Dysgeusia (Nervous system disorders) | 5 (5)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5)
Hemoglobinuria (Renal and urinary disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 7 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (9)
Neutrophil Count Decreased (Investigations) | 4 (4)
Constipation (Gastrointestinal disorders) | 7 (8)
Glucose Intolerance (Metabolism and nutrition disorders) | 1 (1)
INR Increased (Investigations) | 1 (1)
Hemoglobin Increased (Investigations) | 2 (3)
Abdominal Pain (Gastrointestinal disorders) | 2 (5)
Diarrhea (Gastrointestinal disorders) | 6 (7)
Flank Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Cholesterol High (Investigations) | 3 (3)
Accessory Nerve Disorder (Nervous system disorders) | 1 (1) — Sensory Soles of Feet
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Nervous System Disorders - Sensory (Nervous system disorders) | 1 (1)
Phosphorus High (Investigations) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
CPK Increased (Investigations) | 1 (1)
Hearing Impaired (Ear and labyrinth disorders) | 5 (6)
Lymphocyte Count Decreased (Investigations) | 2 (3)
Depression (Psychiatric disorders) | 2 (3)
Palmar-Plantar Erythrodysesthesia Syndrome (Musculoskeletal and connective tissue disorders) | 2 (2)
Bladder Spasm (Renal and urinary disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Urinary Tract Pain (Renal and urinary disorders) | 1 (2)
Paresthesia (Nervous system disorders) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 3 (4)
Dry Mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Gait Disturbance (General disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (3)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2 (2)
Dehydration (Social circumstances) | 1 (1)
Weight Loss (Investigations) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 1 (2)
Alanine Aminotransferase Increased (Investigations) | 1 (2)
Hepatobiliary Disorders (Hepatobiliary disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 1 (1)
Vaginal Infection (Infections and infestations) | 1 (3)
Skin Infection (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Thromboembolic Event (Vascular disorders) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 11 (22)
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle Weakness Left-Sided (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes